CLINICAL TRIAL: NCT02828176
Title: Hemodynamics Effects of Left Lateral Tilt on the Full Term Pregnant Females
Brief Title: The Effect of Left Uterine Displacement on Parturient Cardiovascular System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cardiometry
Record Dates: First submitted 2016-06-21; First posted 2016-07-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cardiac Output
Keywords: cardiometry; uterine displacement
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: electric cardiometry — The following measured variables were recorded using electric cardiometry heart rate, stroke volume, cardiac output, systemic vascular resistance.
  these parameters are measured on arrival to operating room before subarachnoid block in three different angles of lateral uterine tilt ( 0, 15 and 30 degrees )
Procedure: IV line insertion — two Iv lines are inserted and 500cc crystalloid is administered to parturient .
Procedure: spinal anesthesia ( subarachnoid block ) — Subarachnoid block (SAB) was performed in sitting position under complete asepsis using 25 g spinal needle. SAB was achieved by intrathecal injection of 10 mg hyperbaric bupivacaine plus 25ug fentanyl. Success of SAB was tested within five minutes after drug injection. SAB was considered successful if adequate block reached T4 dermatome.
Procedure: electric cardiometry — after SAB the following measured variables were recorded using electric cardiometry heart rate, stroke volume, cardiac output, systemic vascular resistance at three different angles of left uterine lilt (0,15,30 degrees)

SUMMARY:
The aim of the study is to investigate the effect of different angles of lateral tilt on the maternal hemodynamics before and after spinal anesthesia

DETAILED DESCRIPTION:
At operating room, patients will be monitored using non invasive blood, ECG, pulse oximeter and electrical cardiometry. Baseline readings will be taken in supine position then repeated after putting the patient in left lateral position with angle 15 then 30 degrees.

Then two IV lines will be inserted and 500cc crystalloid will be administered. Subarachnoid block will be performed in sitting position under complete aseptic conditions using 25 g spinal needle. Subarachnoid block will be achieved by injecting 10 mg hyperbaric bupivacaine plus 25 ug fentanyl. The block will be considered successful if adequate block reached T4 dermatome.

After successful block the hemodynamic variables will be recorded in the same positions as before (0,15, 30 degrees left uterine tilt).

A minimum number of 61 patients was calculated to have a study power of 80% and alpha error of 0.05.

SPSS Chicago 18 software will be used for data analysis. Categorical data will be presented as frequencies, continuous variables will presented as mean ± standard deviation and will be analyzed using on way analysis of variance (ANOVA) with post-hoc pairwise comparisons using bonferroni test. A P value of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* full term, singleton, American society of anesthesiologists (ASA) I and II pregnant women scheduled for cs

Exclusion Criteria:

* BMI > 35 Kg/m2
* polyhydramnios
* history of impaired cardiac contractility
* valvular heart disease
* cardiac arrhythmias
* hypertensive pregnancy disorders
* fetal abnormalities

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
change in cardiac output (L/min) before anesthesia | baseline : 5min after putting the patient in supine position then 1min after left uterine tilt at 15 and 30 degrees
  measured by electric cardiometry (ICON; Cardiotonic, Osypka; Berlin, Germany).
change in cardiac output (L/min) after spinal anesthesia | baseline after assessing adequate block reaching T4 dermatome then 1 min after left uterine tilt at 15 and 30 degrees
  measured by electric cardiometry (ICON; Cardiotonic, Osypka; Berlin, Germany).

SECONDARY OUTCOMES:
change in systemic vascular resistance (dyn.s/cm5) | baseline : 5min after putting the patient in supine position ( at 0, 15, 30 left uterine tilt ). Then 1 min after assuring adequate level of spinal block
change in mean arterial blood pressure (mmHg) | baseline : 5min after putting the patient in supine position ( at 0, 15, 30 left uterine tilt ). Then 1 min after assuring adequate level of spinal block
  measured by oscillometry in mmHg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] HOWARD BK, GOODSON JH, MENGERT WF. Supine hypotensive syndrome in late pregnancy. Obstet Gynecol. 1953 Apr;1(4):371-7. No abstract available. PMID 13055188
- [Background] Higuchi H, Takagi S, Zhang K, Furui I, Ozaki M. Effect of lateral tilt angle on the volume of the abdominal aorta and inferior vena cava in pregnant and nonpregnant women determined by magnetic resonance imaging. Anesthesiology. 2015 Feb;122(2):286-93. doi: 10.1097/ALN.0000000000000553. PMID 25603203
- [Background] Cluver C, Novikova N, Hofmeyr GJ, Hall DR. Maternal position during caesarean section for preventing maternal and neonatal complications. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD007623. doi: 10.1002/14651858.CD007623.pub3. PMID 23543552
- [Derived] Hasanin A, Soryal R, Kaddah T, Raouf SA, Abdelwahab Y, Elshafaei K, Elsayad M, Abdelhamid B, Fouad R, Mahmoud D, Hassabelnaby Y. Hemodynamic effects of lateral tilt before and after spinal anesthesia during cesarean delivery: an observational study. BMC Anesthesiol. 2018 Jan 15;18(1):8. doi: 10.1186/s12871-018-0473-0. PMID 29334907